CLINICAL TRIAL: NCT07115407
Title: External Validation of the POGO Score for Classification of Videolaryngoscopic Intubation in Children and Comparison With the Quality of the Glottic View Rated on Visual Analogue Scales - Post-hoc Analysis of the Prospective PeDiAC Study
Brief Title: Validation of the POGO Score for Classification of Videolaryngoscopy in Children - Post-hoc Analysis of the PeDiAC Study
Acronym: POGO-KIDS
Status: Active, not recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-300614-WF
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Intubation, Pediatric; Intubation; Difficult or Failed; Airway Management; Airway Complication of Anesthesia
Keywords: POGO score; Pediatric airway management; Videolaryngoscopic intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has been assumed that the percentage of glottic opening (POGO) score might enhance the classification of videolaryngoscopic tracheal intubation by offering a more objective rating of glottic exposure but studies in children are lacking. This post hoc analysis of the prospective observational PeDiAC study aims to investigate, if classifying difficult videolaryngoscopic tracheal intubation with the POGO score is superior to a subjective rating of the quality of the glottic view on visual analogue scales (VAS). Post hoc video analysis will be performed by multiple independent raters. A secondary aim is to determine the diagnostic performance of the POGO and VAS for the prediction of relevant user- and patient-centered outcomes and to assess the inter-rater reliability of the POGO score.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing general anesthesia with tracheal intubation in the study center
* Informed consent obtained
* Age < 18 years

Exclusion Criteria:

* Anesthetist prefers conventional laryngoscopy
* Indication for intubation via a bronchoscope or awake intubation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Consecutive sampling: Pediatric patients undergoing general anesthesia with videolaryngoscopic tracheal intubation in the study center
Sampling Method: Non-Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Difficult videolaryngoscopic intubation | 1 hour
  Defined as a difficult airway alert issued by the airway operator following videolaryngoscopy

SECONDARY OUTCOMES:
Multiple laryngoscopy attempts | 1 hour
  More than one laryngoscopy attempt required until airway established
Multiple tracheal intubation attempts | 1 hour
  More than one tracheal intubation attempt until airway established
First attempt success rate | 1 hour
  Percentage of successful intubations with one attempt at laryngoscopy and intubation
Percentage of glottic opening (POGO) score | 1 hour
  Best glottic view obtained during videolaryngoscopy assessed with the POGO score (%)
Quality of glottic visualization | 1 hour
  Subjective ratings on visual analog scales (0 to 100; higher values indicate better glottic view)
Tracheal intubation time | 1 hour
  Time until successful tracheal intubation
Airway-related adverse events | 1 hour
  Laryngospasm; bronchospasm; airway, oral, soft tissue or dental trauma; laryngeal swelling or use of corticosteroids to reduce swelling risk; oesophageal intubation; pulmonary aspiration; and severe hypoxaemia
Difficulty of videolaryngoscopic tracheal intubation | 1 hour
  Difficulty of videolaryngoscopic tracheal intubation assessed by the PeDiAC score (0-8; higher values indicate increased difficulty)
Severe hypoxaemia | 1 hour
  Oxygen saturation < 70% or hypoxaemia-related bradycardia
Prolonged tracheal intubation | 1 hour
  Tracheal intubation time > 90 sec

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center for Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany